CLINICAL TRIAL: NCT02729259
Title: Water Friendly Virtual Reality for Burns
Brief Title: H2O VR for Burns 2015
Acronym: H2OWC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of General Medical Sciences (NIGMS) (NIH)
Collaborators: University of Washington (Other)
Responsible Party: Principal Investigator, David R. Patterson, Professor, National Institute of General Medical Sciences (NIGMS)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 50416EB/002594
Record Dates: First submitted 2016-03-31; First posted 2016-04-06 (Estimated); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Pain; Burn
Keywords: VRD
MeSH Terms: conditions — Pain; Burns

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- Virtual Reality Snowworld (Other): The subjects will receive Virtual Reality Distraction (VRD) during their wound care procedure. The nurse will be doing their wound care.
  Interventions: Behavioral: Virtual Reality Snowworld
- Virtual Reality slides of nature (Other): The subjects will see several slides of the nature through virtual reality goggles during their wound care. The nurse will be doing the wound care.
  Interventions: Behavioral: Virtual Reality slides of nature
- Control standard nurse wound care (Other): The subjects will receive their standard care during wound care. The nurse will be doing the wound care.
  Interventions: Behavioral: Control standard nurse wound care

INTERVENTIONS:
Behavioral: Virtual Reality Snowworld — The subjects will receive Virtual Reality Snowworld during their wound care procedure. The nurse will be doing their wound care.
  Arms: Virtual Reality Snowworld
Behavioral: Virtual Reality slides of nature — The subjects will receive Virtual Reality Slides of Nature during their wound care procedure. The nurse will be doing their wound care.
  Arms: Virtual Reality slides of nature
Behavioral: Control standard nurse wound care — The subjects will receive their standard care during wound care. The nurse will be doing the wound care.
  Arms: Control standard nurse wound care

SUMMARY:
This study is designed to find additional methods to reduce pain during wound care. In this study the investigators use virtual reality (a form of distraction) in addition to pain medication during a burn wound care.

DETAILED DESCRIPTION:
This study will employ a randomized within-subjects design. There are three different conditions in this study. By randomization, the participants will experience at least two of the conditions and likely all three, depending on the number of their wound care sessions. All subjects will always receive all their usual pain medications for all treatment conditions. The three conditions are: High Tech Virtual Reality (VRD), Low Tech Virtual Reality (Nature Slides), and standard wound care (no VR). The subjects will be randomly assigned to receive some portions of their wound care sessions during High Tech Virtual Reality (VRD), some portions during Low Tech Virtual Reality (Nature Slides), and some portions with standard wound care, no virtual reality. The treatment orders will be randomized. After each treatment condition the investigators will ask subjects one pain question about their pain intensity during the most recent treatment condition.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* Compliant and able to complete questionnaires
* No history of psychiatric disorder
* Not demonstrating delirium, psychosis or any form of Organic Brain Disorder
* Able to communicate verbally
* English-speaking

Exclusion Criteria:

* Age less than 18 years
* Not capable of indicating pain intensity
* Not capable of filling out study measures
* Evidence of traumatic brain injury
* History of psychiatric disorder
* Demonstrating delirium, psychosis or any form of Organic Brain Disorder and associated memory problems
* Unable to communicate orally
* Receiving prophylaxis for alcohol or drug withdrawal
* Developmental disability
* Any face/head/neck injuries that interfere with the use of Virtual Reality equipment
* Non-English Speaking
* Extreme susceptibility to motion sickness
* Seizure history

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
"Pain and anxiety" as measured by Graphic Rating Scale | up to an hour
  Pain and anxiety is being measured

CONTACTS AND LOCATIONS:
Overall Officials: David R. Patterson, Ph.D., Principal Investigator — University of Washington
Locations (1):
- Harborview Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No